CLINICAL TRIAL: NCT05894746
Title: GFREE - A Study for Improved Blood Sugar Levels, Reduced Inflammation and for Increasing Knowledge of the Connection Between Diabetes and COVID-19.
Brief Title: Gfree - For Improved Blood Sugar and Reduced Inflammation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: University of Skövde (Other); Sahlgrenska University Hospital (Other); Ekhaga foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GFREE
Record Dates: First submitted 2023-05-05; First posted 2023-06-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; Celiac Disease; Autoimmunity; Metabolic Disease
Keywords: gluten; probiotics; diet
MeSH Terms: conditions — Diabetes Mellitus; Celiac Disease; Autoimmune Diseases; Metabolic Diseases | interventions — Diet, Gluten-Free; Probiotics; Glutens

STUDY DESIGN:
Intervention Model Description: Four week crossover trial with three arms, gluten-free, gluten and gluten with probiotic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- gluten-free (Experimental): The study participants will start the gluten-free diet and be asked to exchange any products they normally buy with similar products. Three days in the week they will eat a meal with gluten free pasta. Two to six hours after the meal they will take samples at home and store until they return to the clinic.
  Interventions: Dietary Supplement: gluten-free
- gluten (Active Comparator): The study participants will continue the gluten-free diet and be asked to exchange any products they normally buy with similar products. Three days however, in the week they will eat a meal with regular gluten containing pasta. Two to six hours after the meal they will take samples at home and store until they return to the clinic.
  Interventions: Dietary Supplement: gluten-free; Dietary Supplement: gluten
- probiotic (Active Comparator): The study participants will continue the gluten-free diet and be asked to exchange any products they normally buy with similar products. During the week they will also take probiotic (Probion, Active) every morning and every evening. Three days however, in the week they will eat a meal with regular gluten containing pasta. Two to six hours after the meal they will take samples at home and store until they return to the clinic.
  Interventions: Dietary Supplement: gluten-free; Dietary Supplement: probiotic

INTERVENTIONS:
Dietary Supplement: gluten-free — see info in arm description
Dietary Supplement: probiotic — see info in arm description
  Arms: probiotic
Dietary Supplement: gluten — see info in arm description
  Arms: gluten

SUMMARY:
The goal of this clinical trial is to reduce inflammation and improve glycemic control in healthy volunteers, parents, as well as children, adolescents and adults with or without diabetes. The main questions it aims to answer are: • does a reduction wheat gluten improve glycemic control and/or inflammatory biomarkers • does a reduction in certain amino acids (which is most common in wheat gluten) improve glycemic control and/or inflammatory biomarkers • can we identify individuals with an inflammatory response, which leads to poor glycemic control. Participants will eat gluten-free products as well as similar products containing gluten. They will also eat gluten together with probiotics to see if an effect of gluten can be reduced. Researchers will compare everyone with themselves (cross-over design) and if possible individuals with and without diabetes.

DETAILED DESCRIPTION:
BACKGROUND AND PURPOSE Many diseases, which are common in high-income countries, have an inflammatory component. In the world's rich countries, about 10% of the population will be diagnosed with a traditional inflammatory autoimmune disease during their lifetime. In an autoimmune disease, the body produces auto-antibodies against the body's own protein and the immune system destroys the body's own tissues. There are hundreds of different types of autoimmune diseases where some of the most common are; celiac disease (gluten intolerance), psoriasis, type 1 diabetes (T1D), multiple sclerosis, rheumatic diseases or thyroid diseases. Diseases such as cardiovascular disease, type 2 diabetes (T2D) and Alzheimer's disease are now also considered to have inflammatory components, and so-called auto-antibodies have been identified that indicate autoimmunity also in these diseases. Autoantibodies have also been identified in COVID-19 patients.

To try to understand the biology behind autoimmunity and inflammatory disease, the investigators have analyzed the entire genome of patients with celiac disease as a model for autoimmunity. Celiac disease is a good so-called model disease for autoimmunity because the autoimmune reaction can be switched on and off with the help of gluten in the diet. With a strict gluten-free diet, virtually all signs of illness disappear and the inflammation ceases. The results from our whole genome analysis showed that genes involved in amino acid signaling were important for disease development and pointed to associations between celiac disease, T2D and anorexia. These results were somewhat surprising and the investigators began to look at the role of nutritional signaling and amino acids in inflammatory processes further.

The purpose of this study is to test whether a reduction in certain amino acids (which is most common in wheat gluten) can improve glycemic control in healthy volunteers, parents, as well as children, adolescents and adults with diabetes and whether levels of inflammatory amino acids may be one of the factors behind the link between diabetes and severe COVID-19 infection.

The participants will, for 4 weeks, eat one week as usual, eat one week wheat gluten-free, one week wheat gluten and one week with gluten and probiotics. The participants will be provided with continuous glucose monitors and activity-tracking bracelets. The investigators will analyze the efficiency of glucose uptake using continuous glucose monitors (CGM). During these four weeks, the research subjects will be admitted for 4 clinical visits (baseline, after 1 week, 2 weeks, 3 weeks) where blood samples will be taken. Also, during these weeks the participant will take capillary blood samples, faeces, urine, buccal swabs and saliva at home and fill out a questionnaire based on diet and risk factors for diabetes and questions about COVID-19.

Total number of participants: 60 Sampling occasions per participant: 15 Follow-up period per participant: 4 weeks Number of years for inclusion: 2 years (20221201-20241201)

ELIGIBILITY:
Inclusion Criteria:

- none

Exclusion Criteria:

- A diagnosis of celiac disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Stabilizing of blood sugar levels | 0 days to 4 weeks
  Continuous glucose monitoring (CGM) data will be analysed together with activity level data, lower glucose peaks after a meal, adjusted for activity level.
Amino acid metabolism | 0 days to 4 weeks
  Lowering of the aminoacid proline

SECONDARY OUTCOMES:
Blood Lipids | 0 days to 4 weeks
  LDL, improved apolipoprotein B (APOB)
Glutathione S Transferases | 0 days to 4 weeks
  Relative Glutathione S Transferases expression levels
Fibrinogen | 0 days to 4 weeks
  Relative Fibrinogen expression levels

OTHER OUTCOMES:
multiomics explorative analyses | 0 days to 4 weeks
  Genomics, transcriptomics2, metabolomics and proteomics analyses are planned

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Torinsson Naluai, PhD, Principal Investigator — Göteborg University; Katarina Ejeskär, PhD, Study Director — University of Skövde
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - University of Skövde, Skövde

IPD SHARING:
Plan to Share IPD: No
No plan at the moment but the aim is to share data as much as possible.